CLINICAL TRIAL: NCT04924582
Title: Learning From Our Patients, Learning From Our Practice: Implementing an Intervention to Support Patients on Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kasey R. Boehmer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-001884
Record Dates: First submitted 2021-06-04; First posted 2021-06-14 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Dialysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capacity Coaching (Experimental): Participants randomized to the Capacity Coaching arm will receive three months of coaching with a Health and Wellness coach. They will receive one one-hour session and five half-hour sessions approximately two weeks apart.
  Interventions: Other: Capacity Coaching
- No Capacity Coaching (No Intervention): Participants randomized to the No Capacity Coaching arm will receive usual care.

INTERVENTIONS:
Other: Capacity Coaching — Capacity Coaching focuses on developing the capacity within patients to adapt, endure, and function optimally in their lives along with illness and treatment.
  Arms: Capacity Coaching

SUMMARY:
The purpose of this research is to gather preliminary estimates of the impact of using Capacity Coaching as an intervention for patients receiving dialysis.

ELIGIBILITY:
Inclusion Criteria:

Clinician Participants:

* Clinicians employed at Mayo Clinic who provide care to patients visiting the Mayo Clinic - Department of Nephrology and Hypertension Dialysis Services.

Patient Participants:

* Adult patients (18 years of age and older).
* Receive long-term dialysis treatment and services at Mayo Clinic.

Exclusion Criteria:

* Minors (under the age of 18 years).
* Non-English speaking.
* Lack the ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Illness Intrusiveness Score at Baseline, 3 Months, 6 Months | Baseline, 3 Months, 6 Months
  The extent to which a person's illness and treatment impact their life. The Illness Intrusiveness Score ranges from 13-91, with a higher score indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kasey R Boehmer, MPH, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials